CLINICAL TRIAL: NCT01775449
Title: Prevention of Oxaliplatin-induced Neuropathic Pain by a Specific Diet
Acronym: NEUROXAPOL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Fondation Apicil (Other); Ligue contre le cancer - Auvergne (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHU-0137; 2011-A00911-40
Record Dates: First submitted 2013-01-07; First posted 2013-01-25 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2016-07

CONDITIONS: Neuropathy; Digestive Cancer System
Keywords: Anticancer drug;; Oxaliplatin;; Digestive cancer system; Acute oxaliplatin-induced hypersensitivity; Hyperalgesia;; Allodynia;; Dysesthesia; Polyamines depleted diet
MeSH Terms: conditions — Digestive System Neoplasms; Hyperalgesia; Paresthesia | interventions — Polyamines

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- polyamines depleted diet (Experimental): • in the group with a polyamines depleted diet : 2-4 cans per day of Polydol® (oral alimentation without polyamines), associated to predefined menus low in polyamines, according to the chemotherapy cycle and for 107 days
  Interventions: Behavioral: Polyamines depleted diet, associating Polydol® cans and predefined menus low in polyamines
- normal polyamines containing diet (Other): • in the control group with a normal polyamines containing diet: 1 can per day of Polydol® associated with predefined menus with normal average in polyamines and for 107 days.
  Interventions: Behavioral: Polyamines depleted diet, associating Polydol® cans and predefined menus low in polyamines

INTERVENTIONS:
Behavioral: Polyamines depleted diet, associating Polydol® cans and predefined menus low in polyamines

SUMMARY:
Use lay language. Oxaliplatin is a reference anticancer drug in the treatment of colorectal cancer. However, its use is hampered by a specific neurotoxicity, which is characterized by acute thermal hypersensitivity, notably to cold temperatures, and by chronic neuropathy appearing with the repetition of chemotherapy cycles.

To this date there is no effective therapy able to prevent and/or to treat these adverse drug reactions. So oncologists are sometimes strained to decrease anticancer doses or to stop chemotherapy; Previously, a polyamine deficient diet has been able to prevent acute oxaliplatin-induced hypersensitivity in animals.

So we hypothesizes that a specific nutritional therapy, a polyamine deprived diet, may prevent acute oxaliplatin-induced hypersensitivity in patients.

DETAILED DESCRIPTION:
This is a prospective, single-center, controlled and interventional study with two parallel groups randomized in single-blind.

After obtaining informed consent, all included patients will be randomized, either:

* in the group with a polyamines depleted diet : 2-4 cans per day of Polydol® (oral alimentation without polyamines), associated to predefined menus low in polyamines, according to the chemotherapy cycle and for 107 days
* in the control group with a normal polyamines containing diet: 1 can per day of Polydol® associated with predefined menus with normal average in polyamines and for 107 days.

Randomization will be performed by considering stratification on the tumor presence or not, because it is one of the polyamines source (Linsalata and Russo, 2008) and could influence the results in the study.

In addition, patient compliance will be collected in the case report form all along the study, and included in the statistical analysis of the study.

ELIGIBILITY:
Inclusion Criteria:

* - Patients affected by gastrointestinal cancer, without cytotoxic neurotoxic chemotherapy, had to receive FOLFOX 4 chemotherapy (folinic acid + 5-FU + oxaliplatin) in the adjuvant, neoadjuvant or palliative situation with an expected period of 8 cures of treatment or 4 months.
* Patients having given their written, free and informed consent
* Patient's members of a social security scheme
* Patients not having participated in another clinical trial within 15 days before its baseline (possibility of participating and / or participate in an observational trial)
* Effective contraception for patients, male or female, in childbearing age.
* Neutrophils > 2.109/L and/or platelet > 100.109/L before the first treatment cycle

Exclusion Criteria:

* - Patient which cannot receive FOLFOX 4 whatever the reason
* Patients < 18 years old and > 70 years old
* Malnourished patient (French National Authority for Health, 2003)
* Patients with all or part of an upper limb amputation
* Diabetic patient
* Patients with neuropathy
* Oral nutrition impossible
* Painful procedures scheduled after the baseline (e.g. surgical excision)
* Neurological disorders (e.g. parkinsonism, stroke ...)
* Alcohol consumption upper 3 alcohol units (30 g) for men and upper 2 alcohol units (20 g) for women
* Patients having already received cytotoxic neurotoxic chemotherapy (taxanes, platinum salts or vinca alkaloids)
* Patients treated for another cancer within 5 years except basal cell skin carcinoma or in situ cervical cancer
* Any unbalanced progressive disease (hepatic failure, renal insufficiency (creatinine clearance <30 mL / min), respiratory failure, congestive heart failure, myocardial infarction within the past 6 months ...)
* Patients requiring Ca2 + or Mg2 + perfusions
* Hypersensitivity or allergy known about one of study product's component
* Pregnant woman or breastfeeding woman
* Legal disability (person deprived of liberty or under guardianship)
* Patients for psychological, social, family or geographical reasons can not be monitored regularly and / or be compliant with the requirements of the study
* Patients already included in another clinical trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-02-02 (Actual); Primary Completion 2015-01-06 (Actual); Study Completion 2015-01-06 (Actual)

PRIMARY OUTCOMES:
Cold pain thresholds | day 42

SECONDARY OUTCOMES:
Cold pain thresholds | day -7, 0, 2, 14, 16, 28, 30, 42, 70, 72, 98, 100, 154
Heat pain thresholds | day -7, 0, 2, 14, 16, 28, 30, 42, 70, 72, 98, 100, 154
DN4 (Douleur Neuropathique en 4 Questions) scores | day -7, 0, 2, 14, 16, 28, 30, 42, 70, 72, 98, 100, 154
HADS (Hospital Anxiety and Depression Scale) score | day -7, 0, 14, 28, 42, 98, 154
Adverse drug reactions (CTCAE (Common Terminology Criteria for Adverse Events)) | day 0, 2, 14, 16, 28, 30, 42, 70, 72, 98, 100, 154
Cancer response | day 154
Oxaliplatin dose intensity | day 154
Erythrocyte polyamine levels | day -7, 0, 14, 28, 42, 70, 98
NPSI ( Neuropathic Pain Symptom Inventory)scores | day -7, 0, 2, 14, 16, 28, 30, 42, 70, 72, 98, 100, 154
QLQ-C30 (Quality of Life questionnaire C30)scores | day -7, 0, 2, 14, 16, 28, 30, 42, 70, 72, 98, 100, 154

CONTACTS AND LOCATIONS:
Overall Officials: Denis PEZET, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Balayssac D, Ferrier J, Pereira B, Gillet B, Petorin C, Vein J, Libert F, Eschalier A, Pezet D. Prevention of oxaliplatin-induced peripheral neuropathy by a polyamine-reduced diet-NEUROXAPOL: protocol of a prospective, randomised, controlled, single-blind and monocentric trial. BMJ Open. 2015 Apr 1;5(4):e007479. doi: 10.1136/bmjopen-2014-007479. PMID 25833669